CLINICAL TRIAL: NCT06226662
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of NM8074 in Patients with Anti-Neutrophil Cytoplasmic Antibody (ANCA)-Associated Vasculitis (AAV)
Brief Title: Study of NM8074 in Patients with Anti-Neutrophil Cytoplasmic Antibody (ANCA)-Associated Vasculitis (AAV)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NovelMed Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NM8074-AAV-501
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be enrolled and stratified in three strata: (1) granulomatosis with polyangiitis (GPA) (2) microscopic polyangiitis (MPA), and (3) renal-limited vasculitis, and then randomized in a 1:1 ratio of NM8074+SOC to Placebo+SOC (6 subjects in each cohort).
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study (subjects and on-site medical/nursing staff at the study site are blinded to study drug/dose assignment). The pharmacy staff preparing the investigational products will not be blinded to NM8074 study drug assignment, but all other site staff, including the Investigator, will be blinded. Unblinding should only be considered for the safety of the subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NM8074 (Experimental): 6 subjects will receive a biweekly dose of 20 mg/kg of NM8074 plus SOC (cyclophosphamide/azathioprine or rituximab plus corticosteroids)
  Interventions: Drug: NM8074
- Placebo (Placebo Comparator): 6 subjects will receive a biweekly dose of placebo plus SOC (cyclophosphamide/azathioprine or rituximab plus corticosteroids)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NM8074 — NM8074 will be administered as an intravenous infusion. In Cohort 1, all subjects will be administered 20 mg/kg of NM8074 intravenously every two weeks for a total of 7 doses from Day 1 to Day 85 of the Treatment Period.
  Arms: NM8074
Drug: Placebo — Saline Placebo will be administered as an intravenous infusion. In Cohort 2, all subjects will be administered saline placebo intravenously every two weeks for a total of 7 doses from Day 1 to Day 85 of the Treatment Period.
  Arms: Placebo

SUMMARY:
This is a Randomized, Double-Blind, Placebo-Controlled Study designed to assess safety, tolerability, and efficacy of NM8074 in AAV patients when used in combination with Standard of Care (SOC) cyclophosphamide/azathioprine or rituximab plus corticosteroids.

DETAILED DESCRIPTION:
The proposed study, NM8074-AAV-501, will initially assign six (6) patients per cohort in a 2-cohort trial. In the first cohort, we will evaluate a biweekly dosing regimen with NM8074 and SOC whereas in the second cohort, we will evaluate placebo with SOC. These studies will assess safety, tolerability, and efficacy of NM8074 in AAV patients when used in combination with SOC cyclophosphamide/azathioprine or rituximab plus corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of granulomatosis with polyangiitis (GPA), microscopic polyangiitis (MPA), or renal limited vasculitis.
* Male and female subjects aged at least 18 years, with newly diagnosed or relapsed Associated Vasculitis (AAV) where treatment with cyclophosphamide or rituximab is needed.
* At least 1 major item, or at least 3 non-major items, or at least the 2 renal items of proteinuria and hematuria on Birmingham Vasculitis Activity Score (BVAS).
* Estimated glomerular filtration rate (eGFR) ≥ 20 mL/ minute.
* Positive ANCA Test: indirect immunofluorescence (IIF) test for P-ANCA or C-ANCA, or positive ELISA test for anti-proteinase-3 (PR3) or anti-myeloperoxidase (MPO) at Screening.
* All patients must be vaccinated prior to dosing with MenACWY Menactra® polysaccharide diphtheria toxoid conjugate vaccination against Neisseria meningitidis serogroups A, C, Y, and W-135. Meningitis B (MenB) meningococcal serogroup B vaccine (Bexsero®) will be administered per local guidelines. If the window of vaccination is short, then patients will be prophylactically treated with appropriate antibiotics. Patients will also be required to have confirmation or administration of vaccination against S. pneumoniae and H. influenzae.
* Willing and able to understand and complete informed consent procedures, including signing and dating the informed consent form (ICF), and complying with the study visit schedule.
* Female partners of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must have a negative pregnancy test at screening and must agree to use highly effective methods of contraception during dosing and for at least 8 weeks after stopping the investigational drug, and for at least 6 months after the last cyclophosphamide dose (if receiving cyclophosphamide) and at least 12 months after the last rituximab dose (if receiving rituximab).
* Male patients and partners of child-bearing potential must agree to use contraceptives and male patients must agree to refrain from donating sperm for the duration of the study.

Exclusion Criteria:

* Severe disease as determined by alveolar hemorrhage, hemoptysis, rapid onset mononeuritis multiplex or central nervous system involvement.
* Patients with rapidly progressive glomerulonephritis
* Any other known multi-system autoimmune disease including eosinophilic granulomatosis with polyangiitis (EGPA, Churg Strauss), systemic lupus erythematosus, Immunoglobulin A (lgA) vasculitis (HenochSchönlein purpura), rheumatoid vasculitis, Sjogren's disease, anti
* glomerular basement membrane disease, or cryoglobulinemia.
* Required dialysis or plasma exchange within 12 weeks prior to screening.
* Have a kidney transplant or disease.
* Received cyclophosphamide within 12 weeks prior to screening; if on azathioprine, mycophenolate mofetil or methotrexate at the time of screening, these drugs must be withdrawn prior to receiving the cyclophosphamide or rituximab dose on Day 1.
* Received intravenous glucocorticoids, >3000 mg methylprednisolone equivalent, within 4 weeks prior to screening.
* Have been taking an oral daily dose of a glucocorticoid of more than 10 mg prednisone-equivalent for more than 6 weeks continuously prior to screening.
* Received rituximab or other B-cell antibody within 52 weeks of screening or 26 weeks provided B cell reconstitution has occurred (i.e., Cluster of Differentiation 19 (CD19) count > 0.01x10^9/L); received anti-tumor necrosis factor (TNF) treatment or other complement inhibitor treatment within 12 weeks prior to screening.
* Currently or previously under other complement inhibitor treatments less than 3 months prior to study Day 1.
* Patients who need the initiation of renal replacement therapy within 7 days
* Have any other clinically significant abnormal laboratory value in the opinion of the investigator.
* History of bone marrow, hematopoietic stem cell, or solid organ transplantation.
* History of currently active primary or secondary immunodeficiency.
* Currently active systemic infection or suspicion of active bacterial, viral, or fungal infection within 2 weeks prior to first dose, or history of unexplained, recurrent bacterial infections.
* Pregnant, planning to become pregnant, or nursing female subjects.
* Females who have a positive pregnancy test result at Screening or on Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving disease response at Day 85 defined as BVAS percent decrease of at least 50% from baseline. | Up to Study Day 85

SECONDARY OUTCOMES:
Number of patients with ANCA positivity (anti-PR3 and anti-MPO) | Up to Study Day 133
Change from Baseline or Percent Change from Baseline in BVAS (Birmingham Vasculitis Activity Score) | Up to Study Day 133
Change from Baseline or Percent Change from Baseline in Vasculitis Damage Index (VDI) | Up to Study Day 133
Change from Baseline or Percent Change from Baseline in C-reactive protein concentration | Up to Study Day 133
Proportion of patients requiring rescue glucocorticoid treatment | Up to Study Day 133
Proportion of patients achieving disease remission on Day 85 defined as BVAS of 0. | Up to Study Day 85
Percent Change from Baseline in urinary Monocyte Chemoattractant Protein-1 (MCP-1):creatinine ratio | Up to Study Day 133
proportion of subject achieving renal response at Day 85 | Up to Study Day 85
  An >20% increase from baseline to Day 85 in eGFR, A >30% decrease from baseline to Day 85 in hematuria, A >30% decrease from baseline to Day 85 in albuminuria
Change from Baseline or Percent Change from Baseline in quality of life (QoL) Assessed via the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale, Version 4. | Up to Study Day 133
  The FACIT-fatigue scale is a 13-item patient-reported measure of fatigue with a 7-day recall period. Items are scored on a 0 - 4 response scale ranging from "Not at all" to "Very much so". All items are summed to create a single fatigue score with a range from 0 to 52 with a better quality of life indicated by a higher score.
Change from Baseline or Percent Change from Baseline in Quality of Life (QoL) Assessed via the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 Scale (QLQ- C30), Version 3.0 | Up to Study Day 133
  All EORTC QLQ-C30 scales and single-item measures range from 0 to 100. This includes 3 symptom scales (fatigue, pain, nausea and vomiting), 5 functional scales (physical, role, cognitive, emotional, and social), single-item questions addressing symptoms like insomnia, dyspnea, loss of appetite, and others that are commonly reported by cancer patients, and the perceived financial impact of the disease. A higher score is associated with a greater quality of life for global health status.
Change from Baseline or Percent Change from Baseline in Quality of Life (QoL) assessed via EQ-5D-5L | Up to Study Day 133
  The EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a self-assessed, health related QoL which measures QoL in a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.
Change from Baseline or Percent Change from Baseline in Quality of Life (QoL) assessed via SF-36v2 | Up to Study Day 133
  The Short Form Health Survey version-2.0 (SF-36v2) questionnaire is a short-form health survey that measures each of the following eight health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Scales are standardized with a scoring algorithm from 0 to 100.

OTHER OUTCOMES:
Change from Baseline or Percent Change from Baseline in Classical Pathway (CP) modulation | Up to Study Day 133
Change from Baseline or Percent Change from Baseline in Factor B levels | Up to Study Day 133
Change from Baseline or Percent Change from Baseline in plasma concentration of NM8074 | Up to Study Day 133
Maximum plasma concentration (Cmax) | Up to Study Day 133
Time corresponding to Cmax (tmax) | Up to Study Day 133
Area under the drug concentration-time curves (AUC0-t) | Up to Study Day 133

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tesar V, Hruskova Z. Complement Inhibition in ANCA-Associated Vasculitis. Front Immunol. 2022 Jul 8;13:888816. doi: 10.3389/fimmu.2022.888816. eCollection 2022. PMID 35880179
- [Background] Xiao H, Hu P, Falk RJ, Jennette JC. Overview of the Pathogenesis of ANCA-Associated Vasculitis. Kidney Dis (Basel). 2016 Mar;1(4):205-15. doi: 10.1159/000442323. Epub 2015 Dec 3. PMID 27536680
- [Background] Chung SA, Langford CA, Maz M, Abril A, Gorelik M, Guyatt G, Archer AM, Conn DL, Full KA, Grayson PC, Ibarra MF, Imundo LF, Kim S, Merkel PA, Rhee RL, Seo P, Stone JH, Sule S, Sundel RP, Vitobaldi OI, Warner A, Byram K, Dua AB, Husainat N, James KE, Kalot MA, Lin YC, Springer JM, Turgunbaev M, Villa-Forte A, Turner AS, Mustafa RA. 2021 American College of Rheumatology/Vasculitis Foundation Guideline for the Management of Antineutrophil Cytoplasmic Antibody-Associated Vasculitis. Arthritis Rheumatol. 2021 Aug;73(8):1366-1383. doi: 10.1002/art.41773. Epub 2021 Jul 8. PMID 34235894
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Glomerular Diseases Work Group. KDIGO 2021 Clinical Practice Guideline for the Management of Glomerular Diseases. Kidney Int. 2021 Oct;100(4S):S1-S276. doi: 10.1016/j.kint.2021.05.021. No abstract available. PMID 34556256
- [Background] Hellmich B, Sanchez-Alamo B, Schirmer JH, Berti A, Blockmans D, Cid MC, Holle JU, Hollinger N, Karadag O, Kronbichler A, Little MA, Luqmani RA, Mahr A, Merkel PA, Mohammad AJ, Monti S, Mukhtyar CB, Musial J, Price-Kuehne F, Segelmark M, Teng YKO, Terrier B, Tomasson G, Vaglio A, Vassilopoulos D, Verhoeven P, Jayne D. EULAR recommendations for the management of ANCA-associated vasculitis: 2022 update. Ann Rheum Dis. 2024 Jan 2;83(1):30-47. doi: 10.1136/ard-2022-223764. PMID 36927642